CLINICAL TRIAL: NCT05143892
Title: Study on Avatrombopag for the Promotion of Platelet Engraftment After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Avatrombopag to Promote Platelet Engraftment After Allo-HSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, HAN Yue, Director of hematology department, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOOCHOW-HY-2021-11
Record Dates: First submitted 2021-11-21; First posted 2021-12-03 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Platelet Disorder
Keywords: Avatrombopag; thrombocytopenia; allogenic hematopoietic stem cell transplantation; engraftment
MeSH Terms: conditions — Blood Platelet Disorders; Thrombocytopenia | interventions — avatrombopag; Palliative Care

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into avatrombopag group or supportive care group at the ratio of 1:1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avatrombopag (Experimental): In the 4-weeks'study,the initial dose of avatrombopag is 20 mg/d. If the patient's PLT count remains less than 20*10^9/L after one week, the maximum dose was increased to 40 mg/d. Avatrombopag will be taken orally with food.
  Interventions: Drug: Avatrombopag
- Supportive care (Other): Patients in this arm receive same treatment as in the avatrombopag group,except any TPO-RAs or recombinant human thrombopoietin.
  Interventions: Other: Supportive care

INTERVENTIONS:
Drug: Avatrombopag — Avatrombopag administered at the described frequency to achieve a target platelet count
  Other Names: Doptelet
  Arms: Avatrombopag
Other: Supportive care — Supportive care other than TPO-RAs or recombinant human thrombopoietin.
  Other Names: support
  Arms: Supportive care

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of avatrombopag for the promotion of platelet engraftment after Allo-HSCT.

DETAILED DESCRIPTION:
Patients with thrombocytopenia (PLT<20×10^9/L) after allogenic hematopoietic stem cell transplantation (Allo-HSCT) who meet Eligibility Criteria were assigned into the avatrombopag group for 4 weeks' treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 18-60 years;
* PLT<20×10^9/L after 14 days of allo-HSCT;
* Expected survival time > 3 months;
* ECOG performance status 0-2;
* Agree to receive the treatment of avatrombopag after Allo-HSCT and must sign the informed consent form.

Exclusion Criteria:

* Pregnant or lactating;
* With severe and uncontrollable infection;
* With graft-versus-host disease (GVHD) with steroid resistance;
* With thrombotic microangiopathy; With active thromboembolism requiring anticoagulation
* With detected disease recurrence due to chimerism by flow cytometry;
* With chronic active hepatitis B and C virus infection;
* With secondary or multiple transplantation, or multiple organ transplantation;
* With severe heart disease, lung disease, diabetes and metabolic diseases;
* HIV positive;
* With a history of PLT dysfunction or bleeding disorders
* With the active hepatic venous occlusion disease, or a history of clinically significant hepatic venous occlusion disease (The disease was defined as the abnormal condition of painful hepatomegaly after transplantation with bilirubin ≥ 6.0 mg/dL);
* With progressive solid tumor;
* With severe bleeding requiring transfusion of more than 2 units of red blood cells, or sudden drop of blood cell volume ≥10% within 7 days prior to screening;
* With any other clinical trial of investigational product or device within 30 days prior to the baseline visit, except for observational study;
* With treatment of thrombopoietin receptor agonist (TPO-RA) one month before enrollment;
* Deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants whose PLT reaches ≥ 20*10^9/L without the need for PLT transfusion. | up to 4 weeks
  Accumulated platelet engraftment ratio

SECONDARY OUTCOMES:
Percentage of participants whose PLT reaches ≥ 50*10^9/L without the need for PLT transfusion. | up to 4 weeks
  Accumulated complete platelet engraftment ratio
The time to achieve PLT ≥ 20*10^9/L without the need of PLT transfusion for consecutive 7 days (Defined as the first day when PLT ≥ 20×10^9/L without relying on platelet transfusion for 7 consecutive days ) | up to 4 weeks
  time duration of platelet engraftment
Volume of PLT transfusion | up to 4 weeks
  Volume of PLT transfusion
Hematopoietic reconstruction condition | up to 4 weeks
  absolute neutrophils, hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Yue Han, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The first affiliated hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou M, Qi J, Gu C, Wang H, Zhang Z, Wu D, Han Y. Avatrombopag for the treatment of thrombocytopenia post hematopoietic stem-cell transplantation. Ther Adv Hematol. 2022 Sep 28;13:20406207221127532. doi: 10.1177/20406207221127532. eCollection 2022. PMID 36185780

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT05143892/Prot_SAP_ICF_000.pdf